CLINICAL TRIAL: NCT00924560
Title: A Multicenter, Open-Label, Randomized, Controlled Study to Compare the Effects on Bone Mineral Density of DR-105 and a 28-Day Cycle Oral Contraceptive Regimen in Healthy, Postmenarchal, Adolescent Females
Brief Title: A Multicenter Study to Evaluate the Effects of a 91-day Oral Contraceptive on Bone Mineral Density in Adolescent Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-105-202
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Bone Mineral Density
Keywords: Adolescents; Bone Mineral Density; Oral Contraceptive
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination; Seasonique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 91-day Levonorgestrel Oral Contraceptive (Experimental): Participants received a 91-day regimen consisting of 84 consecutive days of active combination tablets containing 150 μg levonorgestrel (LNG)/30 μg ethinyl estradiol (EE), followed by 7 days of 10 μg EE tablets for a total of 52 weeks (4 consecutive 91-day cycles).
  Interventions: Drug: 91-day Levonorgestrel Oral Contraceptive
- 28-day Levonorgestrel Oral Contraceptive (Active Comparator): Participants received a 28-day regimen consisting of 21 consecutive days of active combination tablets containing 100 μg LNG/20 μg EE followed by 7 days of placebo tablets for a total of 52 weeks (13 consecutive 28-day cycles).
  Interventions: Drug: 28-day Levonorgestrel Oral Contraceptive
- Untreated Control (No Intervention): Participants received no oral contraceptives during the study.

INTERVENTIONS:
Drug: 91-day Levonorgestrel Oral Contraceptive — Levonorgestrel/ethinyl estradiol 0.15/0.03 mg and ethinyl estradiol 0.01 mg tablet.
  Take 1 tablet daily
  Other Names: levonorgestrel/ethinyl estradiol; DR-105; Seasonique®
  Arms: 91-day Levonorgestrel Oral Contraceptive
Drug: 28-day Levonorgestrel Oral Contraceptive — Levonorgestrel/ethinyl estradiol 0.10/0.02 mg tablet and placebo. Take 1 tablet daily
  Other Names: levonorgestrel/ethinyl estradiol; Lessina®
  Arms: 28-day Levonorgestrel Oral Contraceptive

SUMMARY:
This study is being conducted to compare the effects of a 91-day oral contraceptive (OC) to a 28-day OC regimen on bone mineral density (BMD) in adolescent females.

DETAILED DESCRIPTION:
Participants will be randomized to either a 91-day OC or a 28-day OC. Participants not seeking hormonal contraception who meet eligibility criteria will serve as a control group. Duration of the study for each study participant will be approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenarchal adolescent female 12-18 years old, non-pregnant, nonlactating
* Regular spontaneous menstrual cycles
* Body mass index (BMI): 18 kg/m² to <30 kg/m², weight < 200 lbs
* Others as dictated by the Food and Drug Administration (FDA)-approved protocol

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* History of previous clinically significant adverse event while taking hormonal contraceptives
* Use of any medication which could significantly interfere with study assessments
* Others as dictated by FDA-approved protocol

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1361 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jen Henrick, Study Chair — Teva GBP
Locations (46):
- United States (46):
  - Teva Investigational Site 007, Phoenix, Arizona
  - Teva Investigational Site 018, Phoenix, Arizona
  - Teva Investigational Site 005, Tucson, Arizona
  - Teva Investigational Site 047, North Little Rock, Arkansas
  - Teva Investigational Site 027, La Mesa, California
  - Teva Investigational Site 040, Los Angeles, California
  - Teva Investigational Site 037, Mountain View, California
  - Teva Investigational Site 013, San Diego, California
  - Teva Investigational Site 017, San Diego, California
  - Teva Investigational Site 025, Torrance, California
  - Teva Investigational Site 022, Washington D.C., District of Columbia
  - Teva Investigational Site 004, Boynton Beach, Florida
  - Teva Investigational Site 008, Clearwater, Florida
  - Teva Investigational Site 026, DeLand, Florida
  - Teva Investigational Site 001, Miami, Florida
  - Teva Investigational Site 003, Miami, Florida
  - Teva Investigational Site 028, Tampa, Florida
  - Teva Investigational Site 041, West Palm Beach, Florida
  - Teva Investigational Site 034, Champaign, Illinois
  - Teva Investigational Site 023, Louisville, Kentucky
  - Teva Investigational Site 021, Baton Rouge, Louisiana
  - Teva Investigational Site 030, St Louis, Missouri
  - Teva Investigational Site 009, Lincoln, Nebraska
  - Teva Investigational Site 010, Lawrenceville, New Jersey
  - Teva Investigational Site 038, Port Jefferson, New York
  - Teva Investigational Site 048, Rochester, New York
  - Teva Investigational Site 002, Durham, North Carolina
  - Teva Investigational Site 043, Kernersville, North Carolina
  - Teva Investigational Site 044, New Bern, North Carolina
  - Teva Investigational Site 020, Raleigh, North Carolina
  - Teva Investigational Site 006, Winston-Salem, North Carolina
  - Teva Investigational Site 033, Cleveland, Ohio
  - Teva Investigational Site 012, Medford, Oregon
  - Teva Investigational Site 035, Pittsburgh, Pennsylvania
  - Teva Investigational Site 039, Pottstown, Pennsylvania
  - Teva Investigational Site 036, Providence, Rhode Island
  - Teva Investigational Site 032, Charleston, South Carolina
  - Teva Investigational Site 024, Columbia, South Carolina
  - Teva Investigational Site 046, Dallas, Texas
  - Teva Investigational Site 031, Houston, Texas
  - Teva Investigational Site 045, Houston, Texas
  - Teva Investigational Site 011, Waco, Texas
  - Teva Investigational Site 015, Salt Lake City, Utah
  - Teva Investigational Site 019, Norfolk, Virginia
  - Teva Investigational Site 014, Seattle, Washington
  - Teva Investigational Site 016, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy, postmenarcheal, adolescent females who were either willing to be randomly assigned to 1 of 2 open-label oral contraceptive (OC) treatment regimens or who were not seeking current treatment with hormonal contraceptives and agreed not to use hormonal contraception throughout the 12-month duration of the study (control group).
Pre-assignment Details: Eligible participants initiating treatment with OCs were randomly assigned to one of the two treatment groups; eligible participants not initiating treatment with hormonal contraceptives were assigned to the untreated control group.
  Twenty-six participants at one clinic were excluded from all analyses as the site was closed due to audit findings.
Groups:
- 91-day Levonorgestrel OC: Participants received a 91-day regimen consisting of 84 consecutive days of active combination tablets containing 150 μg levonorgestrel (LNG)/30 μg ethinyl estradiol (EE), followed by 7 days of 10 μg EE tablets for a total of 52 weeks (4 consecutive 91-day cycles).
- 28-day Levonorgestrel OC: Participants received a 28-day regimen consisting of 21 consecutive days of active combination tablets containing 100 μg LNG/20 μg EE followed by 7 days of placebo tablets for a total of 52 weeks (13 consecutive 28-day cycles).
Period: Overall Study
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Started | 458 | 448 | 455
Received Treatment | 422 (Excludes 7 participants at 1 site that was closed. One participant received 28-day OC in error.) | 411 (Excludes 9 participants from one site that was closed due to audit findings.) | 0
Completed | 247 | 240 | 372
Not Completed | 211 | 208 | 83
Not completed — Did Not Meet Protocol Requirements | 4 | 2 | 1
Not completed — Non Compliance with the Protocol | 20 | 15 | 4
Not completed — Physician Decision | 2 | 3 | 4
Not completed — Withdrawal by Subject | 50 | 44 | 18
Not completed — Adverse Event | 39 | 33 | 0
Not completed — Pregnancy | 5 | 7 | 1
Not completed — Lost to Follow-up | 78 | 94 | 45
Not completed — Miscellaneous Reasons | 13 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control | Total
Number analyzed (Participants) | 458 | 448 | 455 | 1361
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (1.61) | 15.9 (1.71) | 14.8 (1.72) | 15.6 (1.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 458 | 448 | 455 | 1361
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 87 | 87 | 72 | 246
  Asian | 3 | 9 | 12 | 24
  Caucasian | 251 | 265 | 255 | 771
  Hispanic | 102 | 79 | 111 | 292
  Other | 15 | 8 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to 12 Months in Lumbar Spine Bone Mineral Density (BMD)
Description: Bone mineral density was measured by dual energy X-ray absorptiometry (DXA) scan. DXA scans were interpreted centrally by blinded, certified technologists.
  Percent change from Baseline was calculated as (BMD at Month 12 - BMD at Baseline)/BMD at Baseline * 100%.
Time Frame: Baseline and Month 12
Population: Per-protocol analysis set, including all participants who received at least 1 dose of study treatment (does not apply to Control group), had both Baseline and one post-baseline assessment via DXA, and who completed all procedures at all scheduled study visits including the 12-month DXA scans, and did not have any major protocol violations.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 238 | 229 | 362
percent change | 2.26 (0.168) | 1.45 (0.171) | 2.50 (0.139)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel OC vs Untreated Control; The primary efficacy endpoint (percent change from baseline to 12 months in lumbar spine BMD) was analyzed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and chronological age, body weight, and Baseline value as covariates; Test type: Non-Inferiority or Equivalence — 91-day levonorgestrel OC was declared to be non-inferior to the untreated control group if the lower bound of the 2-sided 95% confidence interval (CI) was greater than -3%; LS Mean Difference = -0.23, 95% CI 2-sided [-0.67 to 0.20] — Difference = OC group minus the untreated control
Statistical Analysis 2: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — 28-day levonorgestrel OC was declared to be non-inferior to the untreated control group if the lower bound of the 2-sided 95% confidence interval (CI) was greater than -3%; LS Mean Difference = -1.05, 95% CI 2-sided [-1.49 to -0.61] — Difference = OC group minus the untreated control

2. Secondary Outcome: Change From Baseline in Lumbar Spine Bone Mineral Density
Description: Bone mineral density was measured by dual energy X-ray absorptiometry (DXA) scan. DXA scans were interpreted centrally by blinded, certified technologists.
Time Frame: Baseline, Month 6 and Month 12
Population: Per-protocol analysis set
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Groups:
- 91-day Levonorgestrel OC: Participants received a 91-day regimen consisting of 84 consecutive days of active combination tablets containing 150 μg LNG/30 μg EE, followed by 7 days of 10 μg EE tablets for a total of 52 weeks (4 consecutive 91-day cycles).
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 238 | 229 | 362
g/cm^2
  Change from Baseline to Month 6 | 0.02 (0.001) | 0.01 (0.001) | 0.01 (0.001)
  Change from Baseline to Month 12 | 0.02 (0.002) | 0.01 (0.002) | 0.03 (0.001)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel OC vs Untreated Control; Comparison of Change from Baseline to Month 6. ANCOVA model with treatment as a fixed effect and chronological age, body weight, and Baseline value as covariates; Test type: Superiority or Other; LS Mean Difference = 0.00, 95% CI 2-sided [-0.00 to 0.01]
Statistical Analysis 2: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.01, 95% CI 2-sided [-0.01 to -0.00]
Statistical Analysis 3: Comparison: 91-day Levonorgestrel OC vs Untreated Control; Comparison of Change from Baseline to Month 12. ANCOVA model with treatment as a fixed effect and chronological age, body weight, and Baseline value as covariates; Test type: Superiority or Other; LS Mean Difference = -0.00, 95% CI 2-sided [-0.01 to 0.00]
Statistical Analysis 4: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -0.01, 95% CI 2-sided [-0.02 to -0.01]

3. Secondary Outcome: Change From Baseline in Lumbar Spine Bone Mineral Content (BMC)
Description: Bone mineral content was measured by dual energy X-ray absorptiometry (DXA) scans and interpreted centrally by blinded, certified technologists.
Time Frame: Baseline, Month 6 and Month 12
Population: Per-protocol analysis set
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 238 | 229 | 362
g
  Change from Baseline to Month 6 | 1.29 (0.095) | 0.69 (0.097) | 1.12 (0.079)
  Change from Baseline to Month 12 | 1.86 (0.120) | 1.20 (0.122) | 1.94 (0.099)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.17, 95% CI 2-sided [-0.08 to 0.42]
Statistical Analysis 2: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean Difference = -0.43, 95% CI 2-sided [-0.68 to -0.18]
Statistical Analysis 3: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -0.07, 95% CI 2-sided [-0.39 to 0.24]
Statistical Analysis 4: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -0.74, 95% CI 2-sided [-1.05 to -0.42]

4. Secondary Outcome: Change From Baseline in Proximal Femur Bone Mineral Density
Description: as for outcome 2
Time Frame: Baseline, Month 6 and Month 12
Population: Per-protocol analysis set with available Baseline proximal femur DXA scans; participants with available proximal femur DXA scans at each time point are indicated by "n".
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 238 | 228 | 362
g/cm^2
  Change from Baseline to Month 6 (n=238, 227, 358) | 0.01 (0.001) | 0.00 (0.001) | 0.01 (0.001)
  Change from Baseline to Month 12 (n=238, 224, 359) | 0.02 (0.002) | 0.01 (0.002) | 0.01 (0.001)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.00, 95% CI 2-sided [0.00 to 0.01]
Statistical Analysis 2: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.00, 95% CI 2-sided [-0.01 to 0.00]
Statistical Analysis 3: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = 0.01, 95% CI 2-sided [0.00 to 0.01]
Statistical Analysis 4: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -0.00, 0.95% CI 2-sided [-0.01 to 0.00]

5. Secondary Outcome: Change From Baseline in Proximal Femur Bone Mineral Content (BMC)
Description: as for outcome 3
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 238 | 228 | 362
g
  Change from Baseline to Month 6 (n=238, 227, 358) | 0.26 (0.059) | 0.09 (0.061) | 0.13 (0.049)
  Change from Baseline to Month 12 (n=238, 224, 359) | 0.59 (0.066) | 0.28 (0.068) | 0.43 (0.055)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS mean Difference = 0.13, 95% CI 2-sided [-0.03 to 0.28]
Statistical Analysis 2: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.04, 95% CI 2-sided [-0.20 to 0.11]
Statistical Analysis 3: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = 0.16, 95% CI 2-sided [-0.01 to 0.34]
Statistical Analysis 4: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -0.14, 95% CI 2-sided [-0.32 to 0.03]

6. Secondary Outcome: Change From Baseline in Total Body Bone Mineral Density
Description: as for outcome 2
Time Frame: Baseline, Month 6 and Month 12
Population: Per-protocol analysis set with Baseline total body DXA scans. Participants with available total body DXA scans at each time point are indicated by "n".
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 130 | 126 | 150
g/cm^2
  Change from Baseline to Month 6 (n=130, 126, 149) | 0.01 (0.001) | 0.01 (0.001) | 0.01 (0.001)
  Change from Baseline to Month 12 (n=130, 126, 150) | 0.01 (0.002) | 0.01 (0.002) | 0.02 (0.001)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.00, 95% CI 2-sided [-0.01 to 0.00]
Statistical Analysis 2: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.00, 95% CI 2-sided [-0.01 to 0.00]
Statistical Analysis 3: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -0.00, 95% CI 2-sided [-0.01 to -0.00]
Statistical Analysis 4: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -0.00, 95% CI 2-sided [-0.01 to -0.00]

7. Secondary Outcome: Change From Baseline in Total Body Bone Mineral Content (BMC)
Description: as for outcome 3
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: g
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 130 | 126 | 150
g
  Change from Baseline to Month 6 (n=130, 126, 149) | 40.77 (6.571) | 38.70 (6.638) | 46.26 (6.231)
  Change from Baseline to Month 12 (n=130, 126, 150) | 72.86 (8.325) | 63.78 (8.409) | 84.95 (7.871)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -5.48, 95% CI 2-sided [-23.57 to 12.61]
Statistical Analysis 2: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -7.55, 95% CI 2-sided [-25.65 to 10.55]
Statistical Analysis 3: Comparison: 91-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -12.09, 95% CI 2-sided [-34.99 to 10.81]
Statistical Analysis 4: Comparison: 28-day Levonorgestrel OC vs Untreated Control; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS Mean Difference = -21.17, 95% CI 2-sided [-44.08 to 1.74]

8. Secondary Outcome: Change From Baseline in Bone-specific Alkaline Phosphatase
Time Frame: Baseline, Month 6 and Month 12
Population: Per protocol analysis set with Baseline data available; participants with available data at each time point are indicated by "n".
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 238 | 227 | 356
µg/L
  Change from Baseline to Month 6 (n=236, 224, 353) | -6.8 (8.31) | -5.9 (7.84) | -6.2 (10.42)
  Change from Baseline to Month 12 (n=235, 225, 347) | -6.9 (8.64) | -6.6 (8.82) | -10.3 (12.49)

9. Secondary Outcome: Change From Baseline in Serum Deoxypyridinoline
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 234 | 227 | 350
nmol/L
  Change from Baseline to Month 6 (n=234, 224, 349) | -0.1 (2.43) | -0.1 (1.95) | 0.1 (2.33)
  Change from Baseline to Month 12 (n=233, 226, 348) | -0.1 (2.21) | 0.1 (2.05) | -0.1 (2.28)

10. Secondary Outcome: Change From Baseline in Serum Osteocalcin
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 238 | 227 | 357
nmol/L
  Change from Baseline to Month 6 (n=236, 224, 354) | -4.8 (7.00) | -3.9 (6.74) | -5.1 (11.94)
  Change from Baseline to Month 12 (n=235, 225, 348) | -4.5 (6.69) | -3.7 (7.19) | -7.1 (11.74)

11. Secondary Outcome: Change From Baseline in Serum Procollagen 1 N-terminal Propeptide
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 238 | 227 | 356
µg/L
  Change from Baseline to Month 6 (n=237, 225, 355) | -49.9 (58.55) | -38.7 (51.14) | -57.8 (92.58)
  Change from Baseline to Month 12 (n=235, 226, 349) | -50.4 (60.20) | -39.8 (55.73) | -86.0 (118.69)

12. Secondary Outcome: Change From Baseline in Serum Type I Collagen N-telopeptide
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nM bone collagen equivalents (BCE)
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 237 | 227 | 357
nM bone collagen equivalents (BCE)
  Change from Baseline to Month 6 (n=235, 224, 356) | -4.8 (9.69) | -3.9 (10.68) | -0.7 (13.60)
  Change from Baseline to Month 12 (n=236, 225, 350) | -4.5 (10.22) | -4.3 (10.71) | -3.1 (12.64)

13. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event was any untoward medical occurrence in a clinical investigation subject participating in the clinical study, and did not necessarily need to have a causal relationship with treatment or the clinical study. The relationship of each adverse event to study treatment or procedures, and the severity and seriousness of each adverse event was judged by the investigator, as described below.
  A severe AE is defined as incapacitating, with inability to perform usual activities.
  A serious adverse event is an adverse event occurring at any dose that resulted in any of the following outcomes or actions:
  * fatal or life-threatening;
  * required or prolonged inpatient hospitalization;
  * resulted in persistent or significant disability/incapacity;
  * congenital anomaly or birth defect;
  * important medical event.
Time Frame: 12 months
Population: The safety analysis set includes data from all randomly assigned participants who received at least 1 dose of study treatment and from all participants enrolled in the control group who had baseline BMD measures via DXA. One participant randomly assigned to 91-day LNG received 21-day LNG instead and is included in the 21-day LNG group for safety.
Measure: Number; unit: participants
Groups:
- 28-day Levonorgestrel OC: Participants received a 28-day regimen consisting of 21 consecutive days of active combination tablets (containing 100 μg LNG/20 μg EE) followed by 7 days of placebo tablets for a total of 52 weeks (13 consecutive 28-day cycles).
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Number analyzed (Participants) | 421 | 412 | 437
participants
  Any adverse event | 252 | 258 | 274
  Severe adverse event | 14 | 20 | 10
  Treat-related adverse event | 100 | 95 | 7
  Deaths | 0 | 0 | 0
  Other serious adverse events | 9 | 12 | 0
  Withdrawn from study due to adverse events | 34 | 33 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Description: The safety analysis set includes data from all randomly assigned participants who received at least 1 dose of study treatment and from all participants enrolled in the control group who had baseline BMD measures via DXA. One participant randomly assigned to 91-day LNG received 21-day LNG instead and is included in the 21-day LNG group for safety.
Arm/Group | 91-day Levonorgestrel OC | 28-day Levonorgestrel OC | Untreated Control
Serious Adverse Events (participants affected / at risk) | 9/421 | 12/412 | 0/437
Other Adverse Events (participants affected / at risk) | 156/421 | 160/412 | 196/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 91-day Levonorgestrel OC (N=421) | 28-day Levonorgestrel OC (N=412) | Untreated Control (N=437)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Serositis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Hepatitis infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 91-day Levonorgestrel OC (N=421) | 28-day Levonorgestrel OC (N=412) | Untreated Control (N=437)
Nausea (Gastrointestinal disorders) | 18 (20) | 25 (28) | 14 (15)
Nasopharyngitis (Infections and infestations) | 35 (46) | 52 (62) | 53 (91)
Upper respiratory tract infection (Infections and infestations) | 30 (44) | 27 (32) | 53 (79)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (17) | 14 (26) | 22 (26)
Headache (Nervous system disorders) | 65 (124) | 69 (120) | 88 (197)
Dysmenorrhoea (Reproductive system and breast disorders) | 20 (31) | 26 (41) | 37 (88)
Metrorrhagia (Reproductive system and breast disorders) | 29 (40) | 14 (21) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 10 (12) | 30 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.